CLINICAL TRIAL: NCT01997268
Title: A Randomized, Double-Blind, Placebo-Controlled 12-Week Study to Determine the Efficacy of EPA+DHA (SC401B) on Hypertriglyceridemia (TG ≥ 500 mg/dL and ≤ 2000 mg/dL)
Brief Title: The Efficacy of EPA+DHA (SC401B) for Lowering Triglyceride Levels (≥ 500 mg/dL)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never initiated. IND placed on Hold
Sponsor: Sancilio and Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-13-009
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Severe Hypertriglyceridemia
Keywords: Dyslipidemia; Hyperlipidemia; Omega-3 Fatty Acids; Metabolic Diseases; TG ≥500 mg/dL and ≤ 2,000 mg/dL
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias; Hyperlipidemias; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo 6 capsules (1.24 g each) daily for 12 weeks
  Interventions: Drug: Placebo
- SC401B 2 capsules (Experimental): SC401B 2 capsules (1.24 g each) + 4 placebo capsules daily for 12 weeks
  Interventions: Drug: SC401B 2 capsules
- SC401B 4 capsules (Experimental): SC401B 4 capsules (1.24 g each) + 2 placebo capsules daily for 12 weeks
  Interventions: Drug: SC401B 4 capsules
- SC401B 6 capsules (Experimental): SC401B 6 capsules (1.24 g each) daily for 12 weeks
  Interventions: Drug: SC401B 6 capsules

INTERVENTIONS:
Drug: Placebo — Corn Oil
  Arms: Placebo
Drug: SC401B 2 capsules
  Arms: SC401B 2 capsules
Drug: SC401B 4 capsules
  Arms: SC401B 4 capsules
Drug: SC401B 6 capsules
  Arms: SC401B 6 capsules

SUMMARY:
The purpose of this study is to investigate the effects of SC401B (ethyl esters of eicosapentaenoic acid [EPA] and docosahexaenoic acid [DHA] 2 (~1260 mg EPA+DHA), 4 (~2520 mg EPA+DHA) or 6 (~3780 mg EPA+DHA) capsules per day in subjects with hypertriglyceridemia (triglyceride [TG] ≥500 mg/dL and ≤ 2,000 mg/dL). SC401B capsules also contain certain surfactants that may aid in the absorption of EPA and DHA. Based on the results of pharmacokinetic studies of healthy human subjects, unlike Lovaza®, EPA and DHA in SC401B are bioavailable in both the fasted and fed states.

The protocol specified primary endpoint is the difference from the placebo group in the percent change in TG concentration from baseline to week 12 for groups receiving 2, 4, or 6 capsules of SC401B per day. The protocol specified secondary endpoints include percent changes from baseline to week 12 for total cholesterol (TC), LDL-cholesterol (LDL-C), HDL-cholesterol (HDL-C), and non-HDL-cholesterol (non-HDL-C). Additional exploratory variables include VLDL-cholesterol (VLDL-C), LDL-cholesterol particle size, apolipoprotein (Apo) A1, Apo B, Apo C-III, and lipoprotein-associated phospholipase A2 (Lp-PLA2).

An additional objective is to determine the tolerability and safety of SC401B 2, 4 and 6 capsules per day for 12 weeks. Adverse events for SC401B and placebo including burping, fishy taste, upset stomach, loose stools, stools with fishy smell or any other self-reported observations will be evaluated. Additional safety measures will include changes in liver enzymes (AST/ALT) occurring from baseline to week 12 for groups receiving 2, 4, and 6 capsules of SC401B and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, age 18 years
* Have a TG level ≥500 mg/dL and ≤2,000 mg
* Have the ability to understand the requirements of the study and be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]) and agree to abide by the study restrictions and return for the required assessments.
* Be normally active and in good health on the basis of medical history.
* Willing to maintain a stable diet and not alter their physical activity level throughout the study.
* Women of childbearing potential must be willing to use accepted birth control methods throughout the study.

Exclusion Criteria:

* Women who are pregnant, planning to become pregnant, or breastfeed during the study period
* History of pancreatitis
* Hemoglobin A1c > 9.5% (subjects with diabetes mellitus will be required to receive stable therapy)
* History of stroke, myocardial infarction, life-threatening arrhythmia, or coronary vascularization within 6 months before screening
* Thyroid-stimulating hormone > 1.5 x upper limit of normal; clinical evidence of hypothyroidism or thyroid hormonal therapy that has not been stable for

  * 6 weeks before screening
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x upper limit of normal
* An unexplained creatine kinase concentration > 3 x upper limit of normal or creatine kinase elevation due to known muscle disease (e.g., polymyositis, mitochondrial dysfunction)
* Blood donation of ≥1 pint within 30 days before screening or plasma donation within 7 days before screening
* The consumption of >2 alcoholic beverages per day after screening; a history of illicit drug use within 1 year before screening
* A history of symptomatic gallstone disease unless treated with cholecystectomy
* Known nephrotic syndrome or >3 g/day proteinuria
* Allergy or intolerance to omega-3 fatty acids, ethyl esters, or fish; known lipoprotein lipase impairment or deficiency or apoC-II deficiency or familial dysbetalipoproteinemia
* History of cancer (other than basal cell carcinoma of the skin) in the past 2 years; and a history or evidence of major and clinically significant disease that could adversely affect the conduct of the study or patient safety.
* Use acetylcholinesterase inhibitors or memantine, in the prior 2 months to screening
* Use of a lipase inhibitor such as Xenical (orlistat)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fasting Serum Triglycerides | 12 weeks
  The primary endpoints are the differences in mean percent changes from baseline to end-of-treatment (12 weeks) in triglyceride levels between placebo and 2, 4, and 6 capsules per day of SC401B.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Principal Investigator — Biofortis Clinical Research, Inc.